CLINICAL TRIAL: NCT01062230
Title: Bone Effect of Bortezomib in Patients With Relapsed/Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual; PI left primary institution
Sponsor: University of Arkansas (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI35813
Record Dates: First submitted 2010-02-02; First posted 2010-02-04 (Estimated); Results first posted 2015-04-06 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Multiple Myeloma
Keywords: Cancer; Hematologic malignancy
MeSH Terms: conditions — Multiple Myeloma; Neoplasms; Hematologic Neoplasms | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Experimental): All participants enrolled.
  Interventions: Drug: Bortezomib (Velcade)

INTERVENTIONS:
Drug: Bortezomib (Velcade) — Bortezomib will be administered as a 3-5 second bolus IV injection at the dose of 0.7 mg/m2 on days 1, 4, 8, and 11 q. 21 days times three cycles.
  Patients will undergo three 21-day cycles.
  Other Names: Velcade

SUMMARY:
The primary aim of this trial is to determine the effect of a short course (i.e., 3 cycles) of low-dose Bortezomib (Velcade) on bone remodeling and on disease progression. The dose of bortezomib used in this trial of 0.7 mg/m2 is the lowest dose which has shown efficacy in the 3 largest monotherapy trials with bortezomib. 17% of patients in the APEX, 9% patients in CREST and 24% in SUMMIT trials were treated with 0.7 mg/m2 dosages. Bortezomib will be given on days 1, 8, 15, 22 over 42 days to reduce the incidence of possible drug related side effects.

OBJECTIVES:

Primary Objective

The primary objective of this study is to:

* To evaluate the effect of Velcade at 0.7 mg/m2 dose on inducing osteoblast activation as measured by ALP and other bone markers in patients with relapsed/refractory myeloma.

Secondary Objectives

The secondary objectives of this study are to:

* To evaluate the association between osteoblastic activation and myeloma response to Velcade.
* To identify predictive factors for Velcade-associated osteoblastic activation.

DETAILED DESCRIPTION:
Multiple myeloma (MM) accounts for approximately 1% of all malignancies and 10% of hematological tumors, representing the second most frequently occurring hematological malignancy in the United States. At any one time, 50,000 people suffer from MM, and approximately 15,000 are diagnosed each year. The median age is approximately 65 years, although occasionally MM occurs in the second decade of life. Myeloma is a disease of neoplastic plasma cells that synthesize abnormal amounts of immunoglobulin or immunoglobulin fragments. Myeloma is the only hematological malignancy associated with bone disease. Myeloma is a B-cell neoplasia characterized by clonal expansion of plasma cells in the bone marrow. It is the most malignant stage of plasma cell dyscrasias, which also include the precursor stages of MGUS and indolent or smoldering myeloma. Myeloma is frequently associated with lytic bone disease that is responsible for the most debilitating manifestations of the disease, including bone pain and fractures.

Bone disease in myeloma results from the activation of osteoclast and suppression of osteoblast activity in the myelomatous bone marrow. Change in bone turnover rates, expressed as increased osteoblastic and osteoclastic activity, precede the progression pf MGUS or smoldering myeloma to overt myeloma by as long as three years.

Treatment with bisphosphonates reduces bone resorption and also to some degree, bone formation, and over the long-term moderately increases bone density. Other approved antiresorptive therapies have been shown to reduce the risk of fracture in osteoporotic women, but none have been shown to restore normal bone mass or strength. As a result, treatments that directly stimulate bone formation may overcome these limitations, increase bone mass, and improve the quality of life of myeloma patients. Bone disease is responsible for the most severe complications associated with multiple myeloma. As treatment and survival of myeloma patients improve, new therapies to improve complications are important and vitally needed VELCADE™ (bortezomib) for Injection is a small molecule proteasome inhibitor developed by Millennium Pharmaceuticals, Inc., (Millennium) as a novel agent to treat human malignancies. VELCADE is currently approved by the United States Food and Drug Administration (US FDA) and it is registered in Europe for the treatment of multiple myeloma patients who have received at least one prior therapy.

The clinical response to bortezomib observed in a 63-year-old woman with multiple myeloma and the parallel increase in alkaline phosphatase (ALP) has led us and other groups to evaluate the correlation between bone anabolism and myeloma response to bortezomib. After similar elevations were noted in patients responding to bortezomib, thalidomide, dexamethasone combination, ALP levels were analysed in two large bortezomib trials (Roodman, 2008). Giuliani and coworkers (2007) found that bortezomib significantly increased the activity of the critical osteoblast transcription factor, RUNX2, in human osteoblast precursors and stimulated bone nodule formation in vitro. Importantly, they found a significant increase in the number of osteoblasts per mm2 of bone tissue and the number of RUNX2 positive osteoblastic cells in marrow biopsies from myeloma patients that responded to bortezomib. Again, the effect on osteoblasts was only seen in patients whose myeloma responded to bortezomib, making it difficult to distinguish if the increase in osteoblast activity was due to the anti-myeloma effects of bortezomib or direct effects on osteoblasts or both. Terpos and colleagues (2006) have reported that bortezomib also decreased DKK1 and RANKL concentrations and normalized bone remodeling indices in the serum of patients with relapsed myeloma. However, the majority of patients that showed an increase in bone formation markers also showed an antitumor response to bortezomib, making it unclear if the stimulatory effects on bone formation were secondary to the effects of bortezomib on myeloma or due to direct effects on osteoblast differentiation After similar elevations were noted in patients responding to bortezomib, thalidomide, dexamethasone combination, ALP levels were analysed in two large bortezomib trials.

We first completed a retrospective analysis of large Phase 3 trials comparing ALP levels in responders (≥PR) vs nonresponders (≤PR) patients.

Data obtained from the APEX Crest and Summit protocols, have shown that a total of 85 myeloma patients were treated with bortezomib at the dose of 0.7 mg/m2 for different reasons with significant antimyeloma efficacy for multiple cycles. This dose (0.7 mg/m2) will be used in this trial to test if the antimyeloma activity of bortezomib is still associated to bone anabolic effect. Data for the APEX, summit, and CREST trials is on file at Millennium Pharmaceuticals.

Given that this study is a continuation of a previous protocol (UARK 2004-22) when at the dose of 1.3 and 1.0 mg/m2 an antimyeloma effect and associated bone formation were observed. This trial will test the effect of 0.7 mg/m2 (which has been shown to be effective on antimyeloma treatment) on bone formation to determine the minimal dose associated to bone effect.

ELIGIBILITY:
Inclusion Criteria:

1. History of histologically documented MM with relapsed or progressive disease after at least one line of prior therapy.
2. Patient has measurable disease in which to capture response, defined as one or more of the following:

   1. Serum M-protein level > 1.0 gm/dl (10.0 g/L) measured by serum protein electrophoresis or immunoglobulin electrophoresis; or
   2. Urinary M-protein excretion > 200 mg/24 hrs; or
   3. Bone marrow plasmacytosis of > 30% by bone marrow aspirate and/or biopsy; or
   4. Serum Free Light Chains (By the Freelite test) > 2X ULN, in the absence of renal failure
   5. Radiographic evidence of disease
3. Performance status of < 2 as per ECOG scale, unless PS of 3-4 based solely on bone pain.
4. Patients must have a platelet count > 100,000/L and an ANC of at least 1,000/μl.
5. Patients must have adequate renal function defined as serum creatinine ≤2.5 mg/dL.
6. Patients must have adequate hepatic function defined as serum transaminases and direct bilirubin < 3 x the upper limit of normal.
7. Male or female adults of at least 18 years of age.
8. Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
9. Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
10. Growth factors are allowed during the study
11. Male subject agrees to use an acceptable method for contraception for the duration of the study.

Exclusion Criteria:

1. Platelet count of <100x 10(9)/L within 14 days before enrollment.
2. Absolute neutrophil count (ANC) <1.0 x 10(9)/L
3. Serum creatinine ≥ 2.5 mg/dL within 14 days before enrollment.
4. Patient has >Grade 2 peripheral neuropathy within 14 days before enrollment.
5. Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (see section 1.4), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
6. Patients with a history of treatment for clinically significant ventricular cardiac arrhythmias.
7. Patient has hypersensitivity to bortezomib, boron or mannitol.
8. Chemotherapy or radiotherapy received within the previous 4 weeks of study enrollment.
9. Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
10. Patient has received other investigational drugs with 14 days before enrollment
11. Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
12. Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
13. POEMS Syndrome
14. Clinically significant hepatic dysfunction as noted by bilirubin or AST > 3 times the upper normal limit or clinically significant concurrent hepatitis.
15. Uncontrolled, active infection
16. Patients that have taken bisphosphonates within 30 days of screening will not be eligible for this trial.
17. Must not have received VELCADE 90 days prior to enrolling in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Zangari, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: All participants enrolled.
  Bortezomib (Velcade): Bortezomib will be administered as a 3-5 second bolus IV injection at the dose of 0.7 mg/m2 on days 1, 4, 8, and 11 q. 21 days times three cycles.
  Patients will undergo three 21-day cycles.
Period: Overall Study
Arm/Group | All Patients
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 6
Age, Continuous [Median (Standard Deviation); unit: Years] | 71 (9.58)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Maximum Percent Change From Baseline in Intact Parathyroid Hormone Levels on Day 1
Description: All patients received 0.7 mg/m2 of bortezomib on days 1, 4, 8 and 11 of a 21 day cycle, for maximum of three cycles for an average of 18 months. Intact Parathyroid hormone was measured in patients with relapsed/refractory myeloma for osteoblast activation. Other bone markers were examined using similar methods.
Time Frame: Baseline and Day 1
Measure: Number; unit: % change
Arm/Group | All Patients
Number analyzed (Participants) | 6
% change
  Subject 1 | 113.5
  Subject 2 | -9.09
  Subject 3 | 30.7
  Subject 4 | -50
  Subject 5 | 93.6
  Subject 6 | -53.5

ADVERSE EVENTS:
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=6)
hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
platelets (Blood and lymphatic system disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Creatinine, Serum (Metabolism and nutrition disorders) | 1 (1)
Low ANC (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
platelets - Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Albumin - hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
hemoglobin (Blood and lymphatic system disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Weak pulse (Cardiac disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Complete data was not received from the primary institution for all six patients enrolled. Data available is represented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No